CLINICAL TRIAL: NCT01751022
Title: Attain Performa(TM) Quadripolar Lead Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Attain Performa(TM)
Record Dates: First submitted 2012-12-03; First posted 2012-12-17 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac pacing; cardiac resynchronization therapy; left ventricular lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Attain Performa LV Lead (Models 4298, 4398, 4598) (Experimental): N/A: single arm study, separate analysis for each lead model (total of 3).
  Interventions: Device: Device: Attain Performa Pacing Lead (along with a standard CRT-D system)

INTERVENTIONS:
Device: Device: Attain Performa Pacing Lead (along with a standard CRT-D system) — Implant and follow-up of study lead, separate analysis for each lead model

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the Medtronic Attain Performa Quadripolar Leads (Model 4298, 4398, and 4598) during and post the implant procedure. This study will also assess the interactions of the Attain Performa leads with the entire Medtronic CRT-D system.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for implant of a CRT-D device and left-heart lead per local indications (In US only this is based on Class I and II indications for CRT-D implant per HRS/ACC/AHA guidelines)
* Patient (or legally authorized representative) has signed and dated the study-specific Consent Form
* Patient is 18 years of age or older, or is of legal age to give informed consent per local and national law
* Patient is expected to remain available for follow-up visits
* Patient understands the study and agrees to comply with study protocol

Exclusion Criteria:

* Patient has a previous LV lead implanted or previous implant attempt within 30 days of enrollment or has ongoing AEs from a previous unsuccessful implant attempt
* Patient has contraindications for standard transvenous cardiac pacing (e.g., mechanical right heart valve)
* Patient has had a heart transplant (Note: Patients waiting for heart transplants are allowed in the study)
* Patient is contraindicated for < 1 mg dexamethasone acetate
* Patient is currently enrolled or planning to participate in a potentially confounding drug or device study during the course of this study. (Note: Co-enrollment in concurrent studies may be allowed provided that documented pre-approval is obtained from Medtronic's study manager)
* Patient has a life expectancy less than 180 days
* Patient with exclusion criteria required by local law (e.g. age, pregnancy, breast feeding, etc.)

  * In US, women of childbearing potential must have a negative pregnancy test 7 days prior to implant to be included
* Patient is unable to tolerate an urgent thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (121):
- United States (67):
  - Glendale, California
  - Riverside, California
  - San Diego, California
  - San Jose, California
  - Standford, California
  - West Hollywood, California
  - Hartford, Connecticut
  - Atlantis, Florida
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Houma, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Saint Louis Park, Minnesota
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Henderson, Nevada
  - Morristown, New Jersey
  - Ridgewood, New Jersey
  - New York, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Wynnewood, Pennsylvania
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - Temple, Texas
  - Burlington, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (5):
  - Randwick, New South Wales
  - Chermside, Queensland
  - Adelaide, South Australia
  - Heidelberg, Victoria
  - Perth, Western Australia
- Austria (2):
  - Graz
  - Linz
- Belgium (2):
  - Genk
  - Yvoir
- Canada (5):
  - Calgary
  - London
  - Montreal
  - Newmarket
  - Québec
- Santiago, Chile
- Denmark (2):
  - Århus N
  - Copenhagen
- Helsinki, Finland
- France (3):
  - Nantes
  - Rennes
  - Rouen
- Germany (6):
  - Bad Rothenfelde
  - Bernau
  - Bielefeld
  - Chemnitz
  - Heidelberg
  - Trier
- Athens, Greece
- Budapest, Hungary
- India (2):
  - Gurgaon, Haryana
  - Dehli
- Ashkelon, Israel
- Italy (3):
  - Bologna
  - Cefalù
  - Rovigo
- Kuala Lumpur, Malaysia
- Netherlands (3):
  - Eindhoven
  - Maastricht
  - Nieuwegein
- Bergen, Norway
- Bucharest, Romania
- Riyadh, Saudi Arabia
- Serbia (3):
  - Belgrade
  - Kamenitz
  - Niš
- Slovakia (2):
  - Bratislava
  - Košice
- Ljublijana, Slovenia
- Cape Town, South Africa
- Madrid, Spain
- Lausanne, Switzerland
- United Kingdom (3):
  - Bournemouth
  - London
  - Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 1202 Intial enrollments; 77 were excluded due to to the following pre-implant events:
  1. unsuccessful cannulation (25)
  2. death (3)
  3. Exit prior to implant attempt (43)
  4. Attain Performa Lead implant not attempted (6)
  Resulting in 1125 subjects with Attain Performa Lead Implant Attempts
Groups:
- Model 4298: Patients with an implant attempt for the Attain Performa Lead Model 4298
- Model 4398: Patients with an implant attempt for the Attain Performa Lead Model 4398
- Model 4598: Patients with an implant attempt for the Attain Performa Lead Model 4598
Period: Overall Study
Arm/Group | Model 4298 | Model 4398 | Model 4598
Started | 499 | 326 | 300
Completed | 443 (6 month visit) | 282 (6 month visit) | 273 (6 month visit)
Not Completed | 56 | 44 | 27

BASELINE CHARACTERISTICS:
Population: Subjects with an attempted Attain Performa LV Lead implant
Groups:
- Attain Performa LV Lead Model 4298: Subjects with an attempted Attain Performa LV Lead Model 4298 implant
- Attain Performa LV Lead Model 4398: Subjects with an attempted Attain Performa LV Lead Model 4398 implant
- Attain Performa LV Lead Model 4598: Subjects with an attempted Attain Performa LV Lead Model 4598 implant
- Total: Total of all reporting groups
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598 | Total
Number analyzed (Participants) | 499 | 326 | 300 | 1125
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11) | 66 (11) | 67 (11) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 93 | 93 | 329
  Male | 356 | 233 | 207 | 796
Race/Ethnicity, Customized [Number; unit: participants]
  Subject/physician chose not to provide information | 14 | 9 | 5 | 28
  Not reportable per local laws or regulations | 30 | 21 | 48 | 99
  American Indian or Alaska Native | 4 | 0 | 5 | 9
  Asian | 7 | 8 | 17 | 32
  Black or African American | 38 | 21 | 17 | 76
  Hispanic or Latino | 18 | 11 | 11 | 40
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  White or Caucasian | 387 | 252 | 197 | 836
  Two or more races | 1 | 3 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 360 | 249 | 152 | 761
  Malaysia | 0 | 1 | 1 | 2
  Greece | 0 | 1 | 0 | 1
  Saudi Arabia | 9 | 6 | 2 | 17
  Austria | 8 | 0 | 2 | 10
  Netherlands | 13 | 1 | 9 | 23
  Slovakia | 4 | 2 | 7 | 13
  Slovenia | 0 | 5 | 3 | 8
  Chile | 12 | 0 | 0 | 12
  France | 0 | 2 | 8 | 10
  Serbia | 0 | 2 | 8 | 10
  Romania | 11 | 0 | 1 | 12
  Hungary | 0 | 3 | 4 | 7
  United Kingdom | 13 | 4 | 14 | 31
  Switzerland | 2 | 1 | 1 | 4
  India | 3 | 3 | 15 | 21
  Spain | 3 | 1 | 0 | 4
  Canada | 17 | 22 | 21 | 60
  Belgium | 3 | 1 | 5 | 9
  Norway | 5 | 0 | 0 | 5
  Finland | 0 | 3 | 1 | 4
  Denmark | 1 | 1 | 8 | 10
  Italy | 8 | 10 | 10 | 28
  South Africa | 3 | 2 | 2 | 7
  Israel | 0 | 2 | 2 | 4
  Australia | 17 | 1 | 5 | 23
  Germany | 7 | 3 | 19 | 29
New York Heart Association Classification (NYHA) [Number; unit: participants] — NYHA Functional Classification is assessed as following. Class I: No limitation of physical activity. Class II:Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Unable to carry on any physical activity without discomfort. For more details see American Heart Association website http://www.heart.org/HEARTORG/Conditions/HeartFailure/AboutHeartFailure/Classes-of-Heart-Failure_UCM_306328_Article.jsp#.V_5rPPkrJD8
  participants
    I | 8 | 4 | 4 | 16
    II | 125 | 94 | 89 | 308
    III | 352 | 216 | 198 | 766
    IV | 14 | 12 | 9 | 35
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 25 (7) | 26 (7) | 27 (7) | 26 (7)
QRS (Electrocardiogram Complex) [Mean (Standard Deviation); unit: ms] | 155 (23) | 156 (24) | 156 (23) | 156 (23)

OUTCOME MEASURES:

1. Primary Outcome: Lead Complication-free Rate at 6 Months
Description: The three Attain Performa LV leads models are evaluated separately. The primary safety objective is listed as following:
  - Model 4298/4398: The Attain Performa Model 4298/4398 lead will be considered safe if the probability of subjects freed of Attain Performa lead-related complications at 6 months post-implant is greater than 87% (i.e., the one-sided 97.5% lower confidence bound must be greater than 87%).
  - Model 4598: The safety performance of the Attain Performa Model 4598 lead will be characterized by summarizing the probability of subjects who are free from Attain Performa LV lead related complications at 6 months.
  The lower boundaries of the 97.5% confidence intervals for the all lead models are greater than the pacing threshold of 87%, thus concluding that the crtiera was met for all lead models.
Time Frame: Implant to 6 months post-implant
Population: Subjects with an attempted Attain Performa LV Lead Model. Results for lead model 4298 comes from its PMA-S Clinical Report Version 1, 27MAR2014; results for lead model 4398 comes from its PMA-S Clinical Report Version 3, 03SEP2014; results for lead model 4598 comes from its PMA-S Clinical Report Version 1, 29AUG2014.
Measure: Number (97.5% Confidence Interval); unit: Survival Probability (%)
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 499 | 326 | 300
Survival Probability (%) | 96.04 [94.30 to 100] | 98.75 [97.55 to 100] | 96.21 [94.04 to 100]

2. Primary Outcome: LV Pacing Capture Thresholds Per Attain Performa Lead Model
Time Frame: 6 months post-implant
Population: Subjects with Attain Performa LV Lead Model implanted and valid pacing thresholds measured at the 6 month follow-up visit. Results for model 4298 comes from its PMA-S Clinical Report Version 1, 27MAR2014; for model 4398 comes from its PMA-S Clinical Report Version 3, 03SEP2014; for model 4598 comes from its PMA-S Clinical Report V. 1, 29AUG2014.
Measure: Mean (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Attain Performa LV Lead Model 4298: Subjects with Attain Performa LV Lead Model 4298 implanted and valid pacing thresholds measured at the 6 month follow-up visit.
- Attain Performa LV Lead Model 4398: Subjects with Attain Performa LV Lead Model 4398 implanted and valid pacing thresholds measured at the 6 month follow-up visit.
- Attain Performa LV Lead Model 4598: Subjects with Attain Performa LV Lead Model 4598 implanted and valid pacing thresholds measured at the 6 month follow-up visit.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 395 | 266 | 266
percentage of participants | 93.92 [91.09 to 100] | 96.24 [93.20 to 100] | 95.86 [92.72 to 100]

3. Secondary Outcome: Percentage of Subjects With Presence of PNS in All LV Lead Pacing Polarities
Description: Percentage of patients with presence of PNS in all LV lead pacing polarities at 8.0 V at 0.5ms performed at 6-month visit.
Time Frame: 6 months post-implant
Population: Subjects with Attain Performa LV Lead implanted and at least 1 valid pacing threshold at any LV lead pacing polarity measured at the 6 month visit. Results for model 4298 comes from its PMA-S Clinical Report V1, 27MAR14; for model 4398 comes from its PMA-S Clinical Report V3, 03SEP14; for model 4598 comes from its PMA-S Clinical Report V1, 29AUG14.
Measure: Number; unit: percentage of participants
Groups:
- Attain Performa LV Lead Model 4298: Subjects with Attain Performa LV Lead Model 4298 implanted and at least one valid pacing threshold at any LV lead pacing polarity measured at the 6 month follow-up visit.
- Attain Performa LV Lead Model 4398: Subjects with Attain Performa LV Lead Model 4398 implanted and at least one valid pacing threshold at any LV lead pacing polarity measured at the 6 month follow-up visit.
- Attain Performa LV Lead Model 4598: Subjects with Attain Performa LV Lead Model 4598 implanted and at least one valid pacing threshold at any LV lead pacing polarity measured at the 6 month.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 395 | 267 | 267
percentage of participants
  LV1-RV COIL | 42.03 | 44.19 | 44.57
  LV1-LV2 | 38.48 | 40.45 | 35.58
  LV1-LV3 | 38.99 | 40.45 | 35.58
  LV1-LV4 | 34.18 | 34.83 | 37.83
  LV2-RV COIL | 33.92 | 33.71 | 27.72
  LV2 -LV1 | 34.94 | 32.21 | 27.34
  LV2-LV3 | 12.66 | 18.35 | 10.86
  LV2-LV4 | 27.85 | 25.47 | 22.47
  LV3-RV COIL | 31.39 | 31.84 | 24.72
  LV3-LV1 | 33.42 | 31.46 | 31.84
  LV3-LV2 | 12.91 | 15.36 | 8.61
  LV3-LV4 | 26.58 | 23.60 | 18.73
  LV4-RV COIL | 21.52 | 17.98 | 19.10
  LV4-LV1 | 26.58 | 24.34 | 24.72
  LV4-LV2 | 21.27 | 20.22 | 17.60
  LV4-LV3 | 20.76 | 19.10 | 16.10

4. Secondary Outcome: Percentage of Subjects With Successful Implant Per Attain Performa Lead Model
Time Frame: Implant up to 1-month post implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Model 4298 | Model 4398 | Model 4598
Number analyzed (Participants) | 499 | 326 | 300
percentage of participants | 97.60 [95.84 to 98.75] | 97.55 [95.22 to 98.93] | 98.00 [95.70 to 99.26]

5. Secondary Outcome: Rate of Overall Acceptable Lead Handling Per Attain Performa Lead Model
Time Frame: Implant up to 1-month post implant
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 499 | 326 | 300
percentage of participants
  Acceptable | 98.00 | 98.47 | 98.67
  Unacceptable | 0.20 | 0.31 | 0.33
  No Response | 1.80 | 1.23 | 1.00

6. Secondary Outcome: Pacing Capture Thresholds at the Final Programmed Pacing Polarity
Time Frame: 6 months post-implant
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Attain Performa LV Lead Model 4398: Subjects with Attain Performa LV Lead Model 4398 implanted and valid pacing thresholds measured at the 6 month follow-up.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 395 | 266 | 266
Volts | 1.06 (0.74) | 1.15 (0.76) | 1.10 (0.79)

7. Secondary Outcome: Implant Related Times Per Attain Performa Lead Model
Time Frame: Implant up to 1-month post implant
Population: Subjects with Attain Performa LV Lead Model successfully implanted. Results for model 4298 comes from its PMA-S Clinical Report Version 1, 27MAR2014; for model 4398 comes from its PMA-S Clinical Report Version 3, 03SEP2014; for model 4598 comes from its PMA-S Clinical Report Version 1, 29AUG2014.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Attain Performa LV Lead Model 4298: Subjects with Attain Performa LV Lead Model 4298 implanted successfully.
- Attain Performa LV Lead Model 4398: Subjects with Attain Performa LV Lead Model 4398 implanted successfully.
- Attain Performa LV Lead Model 4598: Subjects with Attain Performa LV Lead Model 4598 implanted successfully.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 487 | 318 | 294
minutes
  Cannulation | 6.3 (9.5) | 8.45 (14.47) | 6.87 (11.19)
  Fluoroscopy | 21.7 (15.4) | 23.00 (17.29) | 18.77 (12.66)
  LV Lead Placement | 13.0 (15.9) | 17.26 (26.21) | 11.82 (14.17)
  Total Operation | 109.6 (49.0) | 107.96 (53.46) | 95.09 (43.38)

8. Secondary Outcome: Pacing Impedance at the Final Programmed Pacing Polarity
Description: Pacing impedance for each LV pacing polarity. Noticed that pacing impedance values are not recorded for reversed LV pacing polarities, since impedance from LV1 to LV2 is the same as from LV2 to LV1.
  Impedance is a measurement of current/resistance between the pacing lead and the cardiac tissue (measured in Ohms).
Time Frame: 6 month post-implant
Population: Subjects with Attain Performa LV lead implanted and complete Medtronic Quad CRT-D system and valid measures of lead impedance at 6-month visit. Results for model 4298 comes from its PMA-S Clinical Report V1, 27MAR14; for model 4398 comes from its PMA-S Clinical Report V3, 03SEP14; for model 4598 comes from its PMA-S Clinical Report V1, 29AUG14.
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- Attain Performa LV Lead Model 4298: Subjects with Attain Performa LV Lead Model 4298 implanted and complete Medtronic Quad CRT-D system and valid measures of lead impedance at 6-month visit.
- Attain Performa LV Lead Model 4398: Subjects with Attain Performa LV Lead Model 4398 implanted and complete Medtronic Quad CRT-D system and valid measures of lead impedance at 6-month visit.
- Attain Performa LV Lead Model 4598: Subjects with Attain Performa LV Lead Model 4598 implanted and complete Medtronic Quad CRT-D system and valid measures of lead impedance at 6-month visit.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 395 | 266 | 267
Ohms
  LV1 to RV Coil | 460.56 (124.26) | 466.24 (123.63) | 496.45 (133.92)
  LV1 to LV2 | 780.49 (228.00) | 802.52 (240.30) | 826.69 (275.82)
  LV1 to LV3 | 776.64 (192.41) | 792.62 (195.78) | 826.15 (278.05)
  LV1 to LV4 | 750.14 (171.98) | 761.79 (175.08) | 799.70 (225.09)
  LV2 to RV Coil | 462.63 (168.82) | 476.71 (193.46) | 483.99 (247.31)
  LV2 to LV3 | 562.40 (179.24) | 568.36 (197.87) | 580.02 (247.99)
  LV2 to LV4 | 730.26 (196.11) | 755.85 (214.04) | 756.48 (257.78)
  LV3 to RV Coil | 450.29 (107.29) | 458.86 (110.62) | 468.90 (247.12)
  LV3 to LV4 | 715.20 (159.58) | 733.30 (164.21) | 740.99 (254.57)
  LV4 to RV Coil | 406.24 (87.12) | 407.17 (87.09) | 421.69 (180.51)

9. Secondary Outcome: Complication Rate for Individual Attain Performa Lead Related Events
Time Frame: 6 month post-Implant
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Number analyzed (Participants) | 487 | 318 | 294
percentage of participants | 3.70 [2.20 to 5.78] | 1.58 [0.51 to 3.64] | 3.74 [1.88 to 6.60]

ADVERSE EVENTS:
Groups:
- Attain Performa LV Lead Model 4298: Subjects with an attempted Attain Performa LV Lead Model 4298 implant. Results as showed in the Model 4298 PMA-S Clinical Report Version 1, 27MAR2014.
- Attain Performa LV Lead Model 4398: Subjects with an attempted Attain Performa LV Lead Model 4398 implant. Results as showed in the Model 4398 PMA-S Clinical Report Version 3, 03SEP2014.
- Attain Performa LV Lead Model 4598: Subjects with an attempted Attain Performa LV Lead Model 4598 implant. Results as showed in the Model 4598 PMA-S Clinical Report Version 1, 29AUG2014.
Arm/Group | Attain Performa LV Lead Model 4298 | Attain Performa LV Lead Model 4398 | Attain Performa LV Lead Model 4598
Serious Adverse Events (participants affected / at risk) | 218/499 | 134/326 | 117/300
Other Adverse Events (participants affected / at risk) | 155/499 | 84/326 | 84/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attain Performa LV Lead Model 4298 (N=499) | Attain Performa LV Lead Model 4398 (N=326) | Attain Performa LV Lead Model 4598 (N=300)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 2 (2)
AFib (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Acute heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Alcoholic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Aortic regurgitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 16 (18) | 12 (16) | 3 (3)
Atrial fibrillation paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 4 (4) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 4 (5) | 5 (7) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atypical angina (Cardiac disorders) | 2 (2) | 2 (9) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disease, unspecified (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 57 (84) | 30 (51) | 33 (46)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Heart fluttering (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac mass (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Monomorphic ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 2 (3) | 3 (3)
Non-ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Permanent atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Persistent atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 4 (4)
Premature ventricular contractions (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Recurrent atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Torsades de pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Unstable angina (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Ventricular ectopic beats (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Ventricular flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 1 (1) | 7 (8)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Benign paroxysmal positional vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Right cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal catastrophe (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1)
Acute duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Antral ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Barrett s esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GI bleed (Gastrointestinal disorders) | 7 (9) | 2 (2) | 2 (2)
GI upset (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastro intestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hernia hiatal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ruptured diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 10 (10) | 7 (24) | 3 (3)
Chest tightness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary restenosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device capturing issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device connection issue (General disorders) | 3 (3) | 2 (2) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug side effect (General disorders) | 0 (0) | 3 (3) | 0 (0)
Elevated pacing threshold (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Implant site hematoma (General disorders) | 2 (2) | 2 (2) | 1 (1)
Implant site pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Inappropriate phrenic nerve stimulation (General disorders) | 1 (1) | 1 (2) | 0 (0)
Inappropriate stimulation of diaphragm (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lead dislodgement (General disorders) | 16 (17) | 3 (4) | 8 (8)
Loss of capture (General disorders) | 1 (1) | 1 (1) | 0 (0)
Multi organ failure (General disorders) | 2 (2) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (4) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Phantom shocks (General disorders) | 0 (0) | 1 (1) | 0 (0)
Premature battery depletion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Substernal chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Undersensing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Unknown cause of death (General disorders) | 4 (4) | 1 (1) | 4 (4)
Weakness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Acute gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
C.difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of toe (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Implant site infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Infection of amputation stump (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 8 (9) | 9 (12)
Prosthesis related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 2 (3) | 1 (1)
Sepsis MRSA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Septic joint (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Sigmoid diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus aureus septicemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcus viridans group infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0) | 2 (2)
Compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Contusion of hip (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Digoxin toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
False aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body in esophagus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured cervical spine (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spurious aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Therapeutic procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Trochanteric femoral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Twiddler s syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Abnormal coagulation profile (Investigations) | 0 (0) | 0 (0) | 1 (1)
Elevated liver enzymes (Investigations) | 1 (1) | 0 (0) | 0 (0)
Subtherapeutic INR (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Volume depletion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Volume overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowel cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CVA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cerebral infarct (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Convulsive seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 2 (2) | 3 (3)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Acute delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (3) | 1 (1)
Acute on chronic renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 5 (6) | 2 (2) | 3 (6)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 2 (3) | 0 (0)
Chronic renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Injury to kidney (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (5) | 1 (1) | 2 (2)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Retention urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Flash pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
AV fistula excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Enterostomy closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial bleeding (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Claudication (Vascular disorders) | 0 (0) | 1 (1) | 1 (3)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension worsened (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive episode (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (6) | 2 (2) | 5 (5)
Ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Leg ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive arteriosclerosis of lower extremities (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral arterial disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Uncontrolled hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attain Performa LV Lead Model 4298 (N=499) | Attain Performa LV Lead Model 4398 (N=326) | Attain Performa LV Lead Model 4598 (N=300)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
AFib (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 12 (13) | 3 (3) | 12 (13)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Atypical angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac sarcoidosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decompensated heart failure (Cardiac disorders) | 31 (35) | 18 (18) | 14 (17)
Junctional rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
LV dyssynchrony (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Monomorphic ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-sustained ventricular tachycardia (Cardiac disorders) | 4 (4) | 2 (2) | 1 (2)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Persistent atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Premature beat atrial (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Recurrent ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (4) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 8 (9) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 8 (11) | 3 (3) | 4 (4)
Chest pressure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device alarm issue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Device connection issue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device damage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device electrical impedance issue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Device migration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device stimulation issue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema extremities (General disorders) | 2 (3) | 0 (0) | 0 (0)
Elevated pacing threshold (General disorders) | 2 (2) | 2 (2) | 1 (1)
Failure to capture (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0)
Impedance increased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site bruising (General disorders) | 2 (2) | 0 (0) | 0 (0)
Implant site burning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site edema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Implant site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Implant site hematoma (General disorders) | 11 (12) | 5 (5) | 0 (0)
Implant site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site numbness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 7 (10) | 4 (6) | 5 (5)
Inappropriate device stimulation of tissue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Inappropriate phrenic nerve stimulation (General disorders) | 18 (20) | 23 (27) | 18 (19)
Inappropriate stimulation of diaphragm (General disorders) | 21 (23) | 13 (14) | 8 (8)
Lead dislodgement (General disorders) | 4 (4) | 0 (0) | 0 (0)
Lead impedance abnormally low (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lead microdislodgement (General disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of capture (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oversensing (General disorders) | 4 (4) | 0 (0) | 2 (2)
Pacing threshold increased (General disorders) | 0 (0) | 3 (3) | 0 (0)
Phantom shocks (General disorders) | 2 (3) | 0 (0) | 0 (0)
Swelling arm (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tissue erosion associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Undersensing (General disorders) | 3 (3) | 0 (0) | 0 (0)
Weakness worsened (General disorders) | 1 (1) | 0 (0) | 0 (0)
Wound healing delayed (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion of chest wall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Coronary sinus dissection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Coronary sinus perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Opiate toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scalp laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation low (Investigations) | 1 (1) | 0 (0) | 0 (0)
Raised blood pressure (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypervolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Volume overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Near syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pre-syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal nocturnal dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme type skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcus cruris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Venous stasis ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial insufficiency peripheral (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0) | 4 (4)
Hypertension worsened (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 11 (14) | 2 (2) | 1 (1)
Low BP (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Superior vena cava stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less